CLINICAL TRIAL: NCT03905980
Title: Evaluation of Risk Factors for Primary Cesarean Section in Egypt
Brief Title: Risk Factors for Primary Cesarean Section in Egypt
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed M Maged, MD, Principal investigator, Cairo University
Other Study IDs: 56
Record Dates: First submitted 2019-04-04; First posted 2019-04-08 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Cesarean Section
MeSH Terms: interventions — Cesarean Section

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Vaginal delivery: woman who terminate their pregnancy by vaginal delivery
  Interventions: Procedure: vaginal delivery
- Cesarean delivery: woman who terminate their pregnancy by cesarean delivery
  Interventions: Procedure: Cesarean section

INTERVENTIONS:
Procedure: vaginal delivery — pregnancy ended by vaginal delivery
  Groups: Vaginal delivery
Procedure: Cesarean section — pregnancy ended by cesarean delivery
  Groups: Cesarean delivery

SUMMARY:
women in their first pregnancy evaluated till delivery for associated risk factors for cesarean delivery

DETAILED DESCRIPTION:
Evaluation of maternal , fetal, delivery place and health care provider rules to determine route of delivery in women during their first pregnancy

ELIGIBILITY:
Inclusion Criteria:

* women in their first pregnancy
* Delivery between 37 and 42 weeks
* Singleton pregnancy _ cephalic presentation

Exclusion Criteria:

* women asked for CS on demand

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: woman carrying their first pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2019-04-30 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
route of delivery in primigravida | at delivery

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, MD, Principal Investigator — Professor
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided